CLINICAL TRIAL: NCT03371147
Title: Patient-Driven Solution in Cancer Care: Improving Outcomes Using a Digital Information and Communication Platform
Brief Title: CancerLife: Patient-Driven Solution in Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: Healthy Platforms, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JWCI-17-1001
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CancerLife (Experimental): Arm A will be asked to download a mobile application called CancerLife. CancerLife is a stand-alone application that is NOT integrated into the patient's electronic health record and will NOT trigger symptom alerts to the treatment team. Participants will be instructed to use the after-visit instructions provided to them by their treatment team for any symptoms or conditions that will require an evaluation by a healthcare provider.
  Interventions: Other: CancerLife
- Usual care (No Intervention): Arm B will receive usual care provided for in the clinics. Usual care may vary between institutions, practices, and providers. Usual care may consist of but is not limited to any combination of the following: history and physical examination, review of systems, distress screening, symptom assessment measures, and/or interval quality of life measures.

INTERVENTIONS:
Other: CancerLife — CancerLife is a patient facing messaging app that gives cancer survivors and caregivers the ability to update family and friends of their health status through their existing social networks and at the same collect psychosocial and symptom reports that can be shared with the patients care team.
  Arms: CancerLife

SUMMARY:
The primary purpose of this study is to evaluate the use of a digital information and communication platform (DICP) in improving outcomes in patients with cancer and their caregivers.

DETAILED DESCRIPTION:
This is a nonblinded, randomized, controlled trial of a digital information and communication platform (DICP) in self-reporting and monitoring of cancer and cancer-treatment related symptoms compared with usual care

Patients initiating and/or receiving systemic treatment for cancer will be enrolled in a nonblinded, randomized, controlled trial of a DICP in self-reporting and monitoring of cancer and cancer-treatment related symptoms compared with usual care. The study will require one (1) study encounter for consenting purposes.

All participants entering their information on the registration page will be contacted by a study team member for informed consent. Eligible subjects who agree to participate in the study and sign the consent form will be will be screened for eligibility. Participants will be randomized 1:1 to two arms:

Arm A will be asked to download a mobile application called CancerLife. CancerLife is a patient facing messaging app that gives cancer survivors and caregivers the ability to update family and friends of their health status through their existing social networks and at the same collect psychosocial and symptom reports that can be shared with the patients care team. Participants will be provided with online or printed instructions on the use of CancerLife and receive a user guide that they can refer on demand. CancerLife is a stand-alone application that is NOT integrated into the patient's electronic health record and will NOT trigger symptom alerts to the treatment team. Participants will be instructed to use the after-visit instructions provided to them by their treatment team for any symptoms or conditions that will require an evaluation by a healthcare provider.

Arm B will receive usual care provided for in the clinics. Usual care may vary between institutions, practices, and providers. Usual care may consist of but is not limited to any combination of the following: history and physical examination, review of systems, distress screening, symptom assessment measures, and/or interval quality of life measures.

Participants in Arm A will be asked to register on CancerLife to start using the broadcasting feature of the app. In addition, they will be asked to complete a series of questions through CancerLife at baseline and every 3 months for up to 2 years. Participants in Arm A will also be asked to complete FACT-G, GAD-7, DST, and QQPPI at those timepoints.

Participants in Arm B will receive usual care provided for in the clinics. They will also be asked to complete the FACT-G, GAD-7, DST, and QQPPI at baseline and every 3 months for up to 2 years..

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of cancer
* Receiving systemic treatment (chemotherapy, biotherapy/immunotherapy, hormonal therapy) that is expected to continue for at least 3 treatment sessions (approximately 9 weeks) from the time of enrollment
* Karnofsky Index ≥50%
* Able to understand and sign informed consent
* Owns and able to use an electronic communication device (smart phone, tablet, laptop, desktop) and answer simple self-report questionnaires on their own

Exclusion Criteria:

* Relevant cognitive impairment
* Participating in a therapeutic clinical trial
* Unable to read and comprehend English language text

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Self-Reported Symptoms | 2 years
  Reduction in severity and occurrence of symptoms

SECONDARY OUTCOMES:
Quality of Life (QOL) | 2 years
  Functional Assessment of Cancer Therapy-General (FACT-G): subscale scores are added to derive total FACT-G score (0-108). The higher the score, the better the QOL.
Anxiety | 2 years
  Generalized Anxiety Disorder 7-item (GAD-7) scale: score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Depression | 2 years
  Depression Screening Tool (DST): score ranges from 0-6, patient with scores of >3 should be further evaluated with other diagnostic instruments.
Emotional state | 2 years
  Tone analyzer and sentiment analysis using IBM Watson
Quality of Physician-Patient Interaction | 2 years
  Questionnaire on the Quality of Physician-Patient Interaction (QQPPI): 14 items with each item ranging from 1-5, higher scores indicating more favorable ratings
Emergency department visits/hospitalizations | 2 years
  Frequency of emergency department visits/hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD PhD, Study Chair — Saint John's Cancer Institute; Marlon G Saria, PhD RN FAAN, Principal Investigator — John Wayne Cancer Institute at Providence Saint John's Health Center
Locations (1):
- John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No